CLINICAL TRIAL: NCT02159417
Title: Feasibility of the Therapeutic Education of the Patients Diabetics Imprisoned at the Paris Jail "La Santé" (Maison d'arrêt Paris La Santé)"
Brief Title: Therapeutic Education of the Patients Diabetics Imprisoned at the Paris Jail
Acronym: EPRIDIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-A00704-41
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Type 1 or 2 Diabetes
Keywords: Evolution of the sport, HbA1C, IMC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Therapeutic Education (Experimental): Intensive training individual or collective teaching
  Interventions: Other: Therapeutic Education

INTERVENTIONS:
Other: Therapeutic Education — Realization of a consultation of educational diagnosis, followed by the participation for every patient to 4 educational collective workshops therapeutic:
  * Knowledge of the disease
  * Food
  * Physical Activity and care of feet
  * The therapeutics
  Other Names: Intensive training individual and collective teaching

SUMMARY:
A lot of data show that therapeutic education is beneficial for diabetic patients. In the French jails, there are very few programs of therapeutic education while this population is usually precarious with no access at care sector before the jail.

The purpose of this study is to determinate if the therapeutic education of the diabetic patients is possible in the Paris jail "La Santé".

DETAILED DESCRIPTION:
The Paris jail "La Santé" welcomes 600 men who stay 5 month on average. Each year, there are between 30 to 40 diabetic patients. In the jail there's a sanitary unit who is a unit of internal medicine of Cochin hospital. This unit includes nurses, pharmacists and medical doctors.

We propose to include in this study all diabetic patients (type 1 and 2) with the realization of a consultation of educational diagnosis, followed by the participation for every patient to 4 educational collective workshops therapeutic (knowledge of the disease, food, physical Activity and care of feet, the therapeutics)

ELIGIBILITY:
Inclusion Criteria:

* Male patient detained in the MAPLS of more than 18 years
* Patient prisoner in the MAPLS for more than 15 days
* Patient follow-up for a diabetes of type 1 or type 2
* Patient informed about the study and not having opposed to this one
* Patient taken out of the disciplinary district which had previously been included for this motive

Exclusion Criteria:

* Patient considered incapable by the investigator to follow an ETP program
* Patient having a bad understanding of the spoken French language
* Patient whose duration of confinement known about the MAPLS is strictly lower than 1 month in the inclusion during the year 2013/2014
* Patient prisoner in the district of isolation
* Patient prisoner in the disciplinary district in the inclusion
* Patient prohibition to communicate with another prisoner already registered on the session to come

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The feasibility of the application of the action ETP in the MAPLS | 3 months
  Rate of participation to at least two therapeutic workshops

SECONDARY OUTCOMES:
Estimation of the satisfaction of the prisoners and the nursing after participation of educational therapeutic workshops | 3 months
  To fill in an auto-questionnaire by means of the scale of Likert in 5 points
biomedical parameters: HbA1c and IMC | 3 months
  Clinical evolution of the patients
The number of hours all in all, for all the activities ETP and by categories of tasks | 3 months
  To evaluate of the mobilized resources
The satisfaction of the staffs as for the implementation and the realization of the experiment | 3 months
  to evaluate of the mobilized resources

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin SILBERMANN, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Laura HARCOUET, Pharm D, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hôpital COCHIN, Paris
  - Maison d'Arrêt Paris La Santé (MAPLS), Paris